CLINICAL TRIAL: NCT04718961
Title: A Phase 2a/2b Randomized Double-Blind Placebo-Controlled Study to Evaluate the Efficacy and Safety of Volixibat in Adult Women With Intrahepatic Cholestasis of Pregnancy and Elevated Serum Bile Acid Concentrations (OHANA).
Brief Title: A Placebo-controlled Study of Volixibat in Subjects With Elevated Serum Bile Acids Associated With Intrahepatic Cholestasis of Pregnancy (OHANA)
Acronym: OHANA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to company's assessment of enrollment feasibility.
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VLX-401; 2020-003448-96 (EudraCT Number)
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: Pruritus; Itch; Itching; Cholestasis; Bile Acid; Pregnancy; Pregnant; Intrahepatic; Liver; ICP
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Pruritus; Cholestasis | interventions — volixibat

STUDY DESIGN:
Intervention Model Description: Randomized Open-label two arm study (Part 1) followed by a randomized double-blind, placebo controlled, study (Part 2)
Who Masked: Participant, Investigator
Masking Description: Masking in Part 2 Only
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Arm 1 - Volixibat 20mg (Experimental): Participants randomized to this arm will receive volixibat 20mg twice daily.
  Interventions: Drug: Volixibat
- Part 1 Arm 2 - Volixibat 80mg (Experimental): Participants randomized to this arm will receive volixibat 80mg twice daily.
  Interventions: Drug: Volixibat
- Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental): Participants randomized to this arm will receive volixibat selected dose (mg) twice daily.
  Interventions: Drug: Volixibat
- Part 2 Arm 2 - Placebo (Placebo Comparator) (Placebo Comparator): Participants in this arm will receive capsules matched to the study drug minus the active volixibat substance, twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Volixibat — Oral capsules, administered twice daily. Volixibat is an ileal bile acid transporter (IBAT) inhibitor.
  Other Names: SHP626
  Arms: Part 1 Arm 1 - Volixibat 20mg; Part 1 Arm 2 - Volixibat 80mg; Part 2 Arm 1 - Volixibat Selected Dose mg
Drug: Placebo — Capsules matched to study drug minus active substance.
  Arms: Part 2 Arm 2 - Placebo (Placebo Comparator)

SUMMARY:
Part 1 is an open-label randomized study of volixibat in patients with Intrahepatic Cholestasis of Pregnancy (ICP) and elevated serum bile acid concentrations (sBA) to evaluate safety and tolerability of two doses of volixibat. Part 2 is a double-blind, placebo controlled, study designed to evaluate the safety and efficacy of a selected volixibat dose.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged ≥18 and ≤45 years with a viable pregnancy.
2. Provide signed informed consent as described in the protocol and willing to comply with all study visits and requirements.
3. Diagnosis of ICP.
4. (Part 2 only) Qualified level of pruritus associated with ICP, during screening.

Exclusion Criteria:

1. At the time of either the screening or baseline visit, decision has already been made to deliver within the next 7 days, for any indication.
2. Known non-reassuring fetal status based upon antepartum testing (e.g., NST/CTG or BPP) at or within 7 days before the baseline visit.
3. Known fetal anomaly likely to result in intrauterine fetal demise or neonatal death within the first 30 days of life.
4. Participating in another ongoing interventional clinical study at screening or planning to participate in another contemporaneous interventional clinical study while participating in this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Yale School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The University of Texas Medical Branch - Galveston, Galveston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- New Zealand (3):
  - Dunedin Hospital, Dunedin, Otago
  - Christchurch Women's Hospital, Christchurch
  - Capital & Coast District Health Board, Wellington Regional Hospital, Wellington
- United Kingdom (10):
  - Medway NHS Foundation Trust, Gillingham, Kent
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - Birmingham Womens and Childrens NHS Foundation Trust, Birmingham
  - University Hospital of Wales, Cardiff
  - St Richard's Hospital, Chichester
  - Barts Health NHS Trust- Whipps Cross University Hospital, London
  - Royal Free London Hospital NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - West Middlesex University Hospital, Middlesex
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

REFERENCES:
- [Derived] Ovadia C, Stone S, Sibai B, Nunes T, Mogul DB, Krishnaswami J, Kahng J, Li F, Warsi QA, Chien E, Vig P, Williamson C. Efficacy, Safety and Tolerability of Volixibat, an IBAT Inhibitor, in Patients With Intrahepatic Cholestasis of Pregnancy. Liver Int. 2026 Mar;46(3):e70523. doi: 10.1111/liv.70523. PMID 41603551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 26 participants were screened at 25 sites in 3 countries (New Zealand, United Kingdom, and United States). Of them, 4 were enrolled in the study.
Pre-assignment Details: After a screening period of up to 10 days during which all procedures listed for the screening visit are completed, eligible patients diagnosed with ICP with screening sBA ≥10 μmol/L during screening or at any time during the current pregnancy were randomized with stratification in a 2-arm (1:1), open-label fashion to receive volixibat 20 mg BID or volixibat 80 mg BID. A total of 26 ICP patients were screened for the study. 22 of these patients were screen failures.
Groups:
- Part 1 Arm 1 - Volixibat 20mg (Experimental): Participants randomized to this arm will receive volixibat 20mg twice daily.
  Volixibat: Oral capsules, administered twice daily. Volixibat is an ileal bile acid transporter (IBAT) inhibitor.
- Part 1 Arm 2 - Volixibat 80mg (Experimental): Participants randomized to this arm will receive volixibat 80mg twice daily.
  Volixibat: Oral capsules, administered twice daily. Volixibat is an ileal bile acid transporter (IBAT) inhibitor.
- Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental): Participants randomized to this arm will receive volixibat selected dose (mg) twice daily.
  Volixibat: Oral capsules, administered twice daily. Volixibat is an ileal bile acid transporter (IBAT) inhibitor.
- Part 2 Arm 2 - Placebo (Placebo Comparator): Participants in this arm will receive capsules matched to the study drug minus the active volixibat substance, twice daily.
  Placebo: Oral capsules, administered twice daily. Capsules matched to study drug minus active substance.
Period: Overall Study
Arm/Group | Part 1 Arm 1 - Volixibat 20mg (Experimental) | Part 1 Arm 2 - Volixibat 80mg (Experimental) | Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental) | Part 2 Arm 2 - Placebo (Placebo Comparator)
Started | 2 | 2 | 0 | 0
Completed | 2 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 2 was early terminated due to lack of enrollment and the company's assessment of enrollment feasibility.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Arm 1 - Volixibat 20mg (Experimental) | Part 1 Arm 2 - Volixibat 80mg (Experimental) | Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental) | Part 2 Arm 2 - Placebo (Placebo Comparator) | Total
Number analyzed (Participants) | 2 | 2 | 0 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 2 | 2 |  |  | 4
  >=65 years | 0 | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 |  |  | 4
  Male | 0 | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 |  |  | 1
  Not Hispanic or Latino | 1 | 2 |  |  | 3
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 |  |  | 0
  White | 1 | 2 |  |  | 3
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 1 | 0 |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 0 |  |  | 1
  United Kingdom | 1 | 2 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Assess the Safety and Tolerability of Volixibat in Participants With ICP
Description: To assess the safety and tolerability of volixibat in participants with ICP on the basis of the following endpoints:
  Proportion of participants experiencing one or more of the following:
  Treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), events of clinical interest (ECIs), and adverse events (AEs) that lead to discontinuation of study drugs.
  Clinically significant laboratory abnormalities
Time Frame: Through to end of treatment, up to 21 weeks
Population: Part 2 was early terminated due to lack of enrollment and the company's assessment of enrollment feasibility.
Measure: Number; unit: participants
Arm/Group | Part 1 Arm 1 - Volixibat 20mg (Experimental) | Part 1 Arm 2 - Volixibat 80mg (Experimental) | Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental) | Part 2 Arm 2 - Placebo (Placebo Comparator)
Number analyzed (Participants) | 2 | 2 | 0 | 0
participants | 2 | 2 |  |

2. Secondary Outcome: Mean Change in the Weekly Average Worst Daily Itch Score as Measured by the Adult Itch Reported Outcome (ItchRO)
Description: Adult Itch Reported Outcome (ItchRO) is a 0 to 10 scale with 0 being "no itch" and 10 being "worst possible itch" where participants are responding to the following question "How would you rate the worst itch you experienced over the last 24hrs?"
Time Frame: Through to end of treatment, up to 21 weeks
Population: Part 2 was early terminated due to lack of enrollment and the company's assessment of enrollment feasibility.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1 Arm 1 - Volixibat 20mg (Experimental) | Part 1 Arm 2 - Volixibat 80mg (Experimental) | Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental) | Part 2 Arm 2 - Placebo (Placebo Comparator)
Number analyzed (Participants) | 2 | 2 | 0 | 0
units on a scale | -2.5 (2.40) | 1.3 (2.31) |  |

3. Secondary Outcome: Proportion of Participants Experiencing One or More of Adverse Perinatal Outcomes
Time Frame: At least one month after delivery.
Population: Part 2 was early terminated due to lack of enrollment and the company's assessment of enrollment feasibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Arm 1 - Volixibat 20mg (Experimental) | Part 1 Arm 2 - Volixibat 80mg (Experimental) | Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental) | Part 2 Arm 2 - Placebo (Placebo Comparator)
Number analyzed (Participants) | 2 | 2 | 0 | 0
Participants | 0 | 2 |  |

ADVERSE EVENTS:
Time Frame: All adverse event data will be collected from first dose of study drug at baseline until whichever of the following time points comes last: 28 days after delivery, or up to 30 days after date of discharge from hospital for mother or for baby, **up to 25 weeks**
Description: Part 2 was early terminated due to lack of enrollment and the company's assessment of enrollment feasibility.
Arm/Group | Part 1 Arm 1 - Volixibat 20mg (Experimental) | Part 1 Arm 2 - Volixibat 80mg (Experimental) | Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental) | Part 2 Arm 2 - Placebo (Placebo Comparator)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Arm 1 - Volixibat 20mg (Experimental) (N=2) | Part 1 Arm 2 - Volixibat 80mg (Experimental) (N=2) | Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental) (N=0) | Part 2 Arm 2 - Placebo (Placebo Comparator) (N=0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Arm 1 - Volixibat 20mg (Experimental) (N=2) | Part 1 Arm 2 - Volixibat 80mg (Experimental) (N=2) | Part 2 Arm 1 - Volixibat Selected Dose mg (Experimental) (N=0) | Part 2 Arm 2 - Placebo (Placebo Comparator) (N=0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | NA | NA
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | NA | NA
Apnoic Episodes (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA | NA — Newborn AE
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | NA | NA
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Headache (Nervous system disorders) | 0 (0) | 1 (1) | NA | NA
Heart Burn (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Intermittent Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA | NA
Intermittent Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA | NA
Intermittent Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA | NA
Mild Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Postnatal Depression (Psychiatric disorders) | 0 (0) | 1 (1) | NA | NA
Premature Labor (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | NA | NA
Raised Blood Pressure (Investigations) | 0 (0) | 1 (1) | NA | NA
Threated Pre-Term Labor (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | NA | NA
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT04718961/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT04718961/SAP_001.pdf